CLINICAL TRIAL: NCT05932706
Title: Intervention Effect of High Definition Transcranial Alternating Current Stimulation (HD-tACS) on Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Director of medical psychological department, Anhui Medical University, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tACS-MDD
Record Dates: First submitted 2023-05-11; First posted 2023-07-06 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2023-06

CONDITIONS: Transcranial Alternating Current Stimulation; Depressive Disorder
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real stimulation (Active Comparator): The central electrode was placed over F3, with return electrodes at Fp1, Fz, F7 and C3. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 15 and 15 seconds, respectively) were applied for 30 minutes per session, twice daily over 7 consecutive days, and the stimulus frequency was set as IAF.
  Interventions: Device: High definition transcranial alternating current stimulation
- sham stimulation (Sham Comparator): In the sham condition, tACS was delivered only during the ramp-up and ramp-down periods (15 and 15 s); no current was delivered during the 30-minute intervention. Participants will receive sham tACS twice daily for two weeks.
  Interventions: Device: sham high definition transcranial alternating current stimulation

INTERVENTIONS:
Device: High definition transcranial alternating current stimulation — tACS is described as a non-invasive form of brain stimulation that uses a low-intensity, alternating current applied directly to the head through scalp electrodes.
  Arms: real stimulation
Device: sham high definition transcranial alternating current stimulation — In the sham condition, tACS was delivered only during the ramp-up and ramp-down periods (15s and 15s); no current was delivered during the 30-minute intervention.
  Arms: sham stimulation

SUMMARY:
To investigate the intervention effect of high definition transcranial alternating current stimulation (HD-tACS) on suicidal ideation in patients with depressive disorder and its underlying neural mechanism by magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
Forty patients with depressive disorder diagnosed by DSM-5 were recruited from the Anhui Mental Health Center and the first affiliated Hospital of Anhui Medical University. All participants underwent a structured interview and routine laboratory examination before and after receiving high definition transcranial alternating current stimulation (HD-tACS) treatment after meeting the inclusion criteria and obtaining informed consent. Each participant will complete the clinical evaluation, magnetic resonance imaging (MRI), electroencephalography (EEG), and HD-tACS treatment conducted by trained researchers at the Anhui Mental Health Center. All the participants were randomized (1:1) to receive an "active HD-tACS" or "sham HD-tACS" treatment protocol. tACS: the central electrode was placed over F3 with return electrodes placed at Fp1, Fz, F7 and C3. Fourteen 2-mA sessions (ramp-up and ramp-down periods of 15 and 15 seconds, respectively) were applied for 30 minutes per session, twice daily over 7 consecutive days, and the stimulus frequency was set as individual alpha frequency (IAF). Sham HD-tACS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 15 and 15 seconds.

Before and after the treatments, the patients received a battery measure of neuropsychological tests, resting EEG, and MRI scans in multimodalities. The neuropsychological assessment included HAMD, MADRS, BDI, HAMA, BSS, C-SSRS, PHQ15, RRS, TEPS, PVAQ, MoCA, Stroop Test, VFT, DST, and AVLT. Multimodal MRI includes 3D-T1, rs-fMRI, and DTI. The symptoms of the patients were followed up one and two months after the end of treatments.

ELIGIBILITY:
Inclusion Criteria:

* the patients were diagnosed by more than 2 psychiatrists and met the diagnostic criteria of DSM-5 for depression, and item 3 of the HAMD≥3.
* the age ranged from 18 to 65 years old, and the length of education was more than 5 years.
* the visual acuity or corrected visual acuity is normal, right-handed, can cooperate with the completion of various experimental tests.

Exclusion Criteria:

* accompanied by severe somatic diseases, such as severe heart, liver, renal insufficiency and so on.
* accompanied by other neurological diseases, such as stroke, epilepsy and so on. pregnant and lactating women.
* accompanied by other mental disorders, such as drug abuse, schizophrenia, schizophrenic affective

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Beck Scale for Suicide Ideation (BSS) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The BSS is a 19-item scale to measure the severity of suicidal ideation, where each item is rated on a scale from 0 to 2. The BSS total score ranges from 0 to 38 with lower scores indicating less suicidal ideation.

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation (BSS) Response Rate (≥50% Improvement From Baseline) | week 1 (end of treatment) and week 5 (end of follow-up)
  The BSS is a self-report measure of suicidal ideation severity, with higher scores indicating greater severity. Response was defined a priori as a 50% or greater reduction in BSS total score from baseline. The BSS response rate was calculated as the proportion of participants meeting this criterion at each postbaseline assessment.
Change in Columbia-Suicide Severity Rating Scale (C-SSRS) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The C-SSRS is a clinician-administered instrument used to assess the severity of suicidal ideation and suicidal behavior. The suicidal ideation module evaluates (1) ideation severity over the past month (rated 1-5, with 0 indicating no suicidal ideation) and (2) ideation intensity across 5 items (eg, frequency and duration), each rated 0-5, yielding a total intensity score ranging from 0 to 25; higher scores indicate more severe suicidal ideation. The suicidal behavior module captures the presence and characteristics of suicidal behaviors (eg, number of attempts and lethality).
Change in Hamilton Depression Rating Scale (HAMD) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The HAMD is a clinician-administered depression assessment and consists of 17 items with a total score range from 0 to 54. A higher score indicates a worse outcome.
Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The MADRS is a 10-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 6. The MADRS total score ranges from 0 to 60, with lower scores indicating less depressive symptoms.
Change in Beck Depression Inventory (BDI) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The BDI is a 13-item scale to measure the severity of depressive episodes, where each item is rated on a scale from 0 to 3. The BDI total score ranges from 0 to 39, with lower scores indicating less depressive symptoms.
Change in Hamilton Anxiety Scale (HAMA) Score | baseline, week 1 (end of treatment), and week 5 (end of follow-up)
  The HAMA is a 14-item scale to measure the severity of anxiety symptoms, where each item is rated on a scale from 0 to 4. The HAMA total score ranges from 0 to 56, with lower scores indicating less anxiety symptoms.
Change in Game of Dice Task (GDT) Score | baseline and week 1 (end of treatment)
  The GDT is a computerized task assessing risk decision-making under explicit probabilities. Participants choose between higher-risk options with lower winning probabilities (<50%) and higher safe options with winning probabilities (≥50%) across 18 trials; outcomes (gains/losses) are presented after each trial. Prespecified outcomes included the number of risky choices, number of safe choices, and a net score (safe choices minus risky choices), with higher net scores indicating safer decision-making.
EEG Measure of Frontal Alpha Asymmetry (FFA) Oscillations | baseline and week 1 (end of treatment)
  EEG recordings were obtained from each subject based on 64 electrode locations of the International 10-20 system (sampling frequency 1000Hz). The change in FFA (8-13 Hz electrical activity) over time was measured.
MRI measures of functional connectivity (FC) | baseline and week 1 (end of treatment)
  the functional connectivity between stimulated target and the whole brain areas; the global and regional activity measures.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghua Tian, PhD, Study Chair — Anhui Medical University
Locations (1):
- Yanghua Tian, Hefei, Anhui, China